CLINICAL TRIAL: NCT03053297
Title: Global PANORAMA Real World Molecular Testing, Treatment Patterns, and Clinical Outcomes in Patients With Locally Advanced or Metastatic NSCLC.
Brief Title: Observational Study of Patients With Locally Advanced or Metastatic NSCLC (Non-Small Cell Lung Cancer)
Acronym: PANORAMA
Status: Terminated | Type: Observational
Why Stopped: Cancelled due to changes in the scientific landscape. Decision was made after thorough evaluation of of pros&cons, ethical as well as regulatory consideration
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160R00010
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: EGFR; EGFR mutation; EGFRm; EGFR-TKI; Health care resource utilization; Health-Related Quality of Life; Locally advanced or metastatic lung cancer; NSCLC; Non-Small Cell Lung Cancer; Observational study; Osimertinib; Personalized medicine; PRO; Patient Reported Outcome; Resistance; T790M; Carcinoma, Non-Small-Cell Lung; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic neoplasms, Neoplasms by site; Lung diseases; Respiratory Tract diseases; Cancer Chemotherapy; Combination Chemotherapy; Immunotherapy; Radiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma, Bronchogenic; Bronchial Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Lung Diseases; Respiratory Tract Diseases | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with EGFR mutation (+) NSCLC: Patients with EGFR mutation-positive locally advanced or metastatic NSCLC who have progressed while on or after receiving front-line EGFR-TKI therapy (e.g., gefitinib, erlotinib, afatinib, or icotinib).
  Interventions: Other: Patient Reported Outcomes
- Patients newly diagnosed NSCLC: Patients newly diagnosed with locally advanced or metastatic NSCLC who are treatment naive or patients who were diagnosed at an earlier stage but have progressed to metastatic NSCLC during the selection period.
  Interventions: Other: Patient Reported Outcomes

INTERVENTIONS:
Other: Patient Reported Outcomes — HRQoL will be assessed using questionnaire EORTC QLQ-C30 and the questionnaire EORTC QLQ-LC 13.
  These two questionnaires are validated instruments, translated in various languages and are not used as an intervention but rather to track patient quality of life and symptom reduction in real-life settings. Data for these patient reported outcomes will be collected prospectively from the time of enrolment until the end of follow-up. The two questionnaires will be self-administered by the patients in both cohorts at the enrolment visit and subsequently every 3 months (±1 month) at routine standard of care scheduled visits. The questionnaires are expected to take about 15 minutes to complete

SUMMARY:
This is an observational cohort study of patients with locally advanced or metastatic NSCLC (non-small cell lung cancer).

Patients will be recruited from participating sites in Europe, Asia, and Canada. The study will include 2 patient cohorts.

DETAILED DESCRIPTION:
Study Design This will be an observational cohort study of patients with locally advanced or metastatic NSCLC (non-small cell lung cancer).

Patients will be recruited from participating sites in Europe, Asia, and Canada. Patients meeting the study inclusion/exclusion criteria will be selected during a 24-month enrolment period per country and will be followed from enrolment in the study until death, loss to follow-up, withdrawal of consent or study end date (whichever occurs earlier). Data Sources Data will be collected following enrolment in the study and entered in the electronic case report form (eCRF). All data will be collected using patient medical records. The investigator will be responsible for ensuring that all the required data is collected and entered into the eCRF. The site will collect the patient questionnaires and the data will be uploaded according to the data entry procedures.

Study Population

* Adult male or female patients (according to age of majority/adulthood as defined by local regulations) who have given written informed consent as per local regulations.
* The primary cohort will include patients with EGFR (epidermal growth factor receptor) mutation-positive locally advanced or metastatic NSCLC who have progressed while on or after receiving front-line EGFR-TKI (tyrosine kinase inhibitors) therapy (e.g., gefitinib, erlotinib, afatinib, or icotinib).
* Additionally, a secondary cohort of patients will include patients newly diagnosed with locally advanced or metastatic NSCLC who are treatment naive or patients who were diagnosed at an earlier stage but have progressed to metastatic NSCLC during the selection period.

Exposures There are no specific drug exposures or interventions being evaluated, as cohort eligibility (for both cohorts) is not exposure-based, but rather disease-based. All molecular testing and treatments will be at the discretion of the treating physician. Study Measures and Outcomes

* Patient demographic and clinical characteristics
* Molecular testing patterns and outcomes
* Treatment patterns
* Physician-reported clinical outcomes
* Cancer-related health care utilization
* Treatment- and biopsy-related complications
* CNS metastases (brain metastases and leptomeningeal metastases) and treatments associated with CNS (central nervous system) metastases
* HRQoL (Health Related Quality of Life) and symptoms Precision and Sample Size Estimations For the primary cohort the minimum sample size recommended for conducting a country-level analysis is 200 patients per country. This is based on the precision estimation calculation for the categorical study measure (% of patients tested) and will allow a maximum of

  * 8.3% precision (i.e., assuming 50% undergoing molecular testing) around the point estimate for the categorical measure. For the secondary cohort the minimum sample size recommended for conducting a country-level analysis is 300 patients which was determined using precision estimates calculated for a categorical (% of patients tested) and a time-to-event (overall survival) measure. The overall study will include approximately 2800-3300 patients across all participating countries across both primary (1200-1300 patients) and secondary (1600-2000 patients) cohorts. Statistical Analysis No formal hypothesis testing is specified. Study measures including patient demographics and clinical characteristics, molecular testing patterns, treatment sequence patterns, physician-reported outcomes (overall survival) and patient-reported outcomes (HRQoL) will be reported by primary and secondary cohorts, unless indicated otherwise. Continuous study measures (e.g., age, duration of therapy) will be reported descriptively with mean, standard deviation, median, minimum and maximum. Frequencies and percentages will be used to document categorical measures of interest (e.g., number and proportion of patients with a post progression molecular test, number and proportion of patients with a T790M mutation) and will include 95% CIs for key outcome variables. Kaplan-Meier curves and median survival will be estimated, overall and on an exploratory basis by clinical and treatment characteristics of interest (provided there are sufficient events available; e.g., chemotherapy vs. targeted therapy) as pre-specified in the statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent - patient consent should be within 6 weeks of index date.
* Adult male or female subjects (according to age of majority/adulthood as defined by local regulations)

Exclusion Criteria:

-Enrolment in studies that prohibit any participation in this non interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Adult male or female patients (according to age of majority/adulthood as defined by local regulations) who have given written informed consent as per local regulations.
  * The primary cohort will include patients with EGFR mutation-positive locally advanced or metastatic NSCLC who have progressed while on or after receiving front-line EGFR-TKI therapy (e.g., gefitinib, erlotinib, afatinib, or icotinib).
  * Additionally, a secondary cohort of patients will include patients newly diagnosed with locally advanced or metastatic NSCLC who are treatment naive or patients who were diagnosed at an earlier stage but have progressed to metastatic NSCLC during the selection period. (In Spain and France the secondary cohort of patient will be limited to patients with EGFR mutation-positive locally advanced or metastatic NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Parameters in the target population associate with molecular testing patters | Patients will be followed from enrolment in the study until death, loss to follow-up, withdrawal of consent or study end date. The minimum follow-up will be 12 months and the maximum allowed follow-up will be 36 months
  * Molecular testing rate defined as the number of patients identified as having received molecular testing divided by the number of patients in the cohorts
  * Changes in testing rates over time (details will be included in the SAP)
  * Molecular testing details including, but not limited to sample type, method of biopsy, testing turnaround time, test type, reason for testing, testing laboratory type, reason for not performing a test
  * Molecular testing results including mutation status and type, test outcome, histologic/phenotypic transformation
Parameters in the target population associate with treatment patterns and associated clinical outcomes | Patients will be followed from enrolment in the study until death, loss to follow-up, withdrawal of consent or study end date. The minimum follow-up will be 12 months and the maximum allowed follow-up will be 36 months
  * Overall survival measured from:
    * the date of initial diagnosis to date of death from any cause to the index date to date of death from any cause (for primary cohort only)
    * the date of first-line treatment until death
    * the date of second-line treatment until death
  * Overall disease progression:
    o from date of treatment initiation until physician-reported progression, initiation of a new cancer-directed line of therapy (proxy for progression), or death
  * For each line of chemotherapy/targeted therapy received:
    * Therapy regimen
    * Therapy duration measured as time from therapy start date to time of therapy end date
    * Number of cycles received
    * Reason for cessation of therapy
    * Time to initiation of new therapy defined as the time from start date of current therapy to start date of subsequent therapy
  * For each surgery or radiotherapy received:
    * Type
    * Site
    * Date
  * Any palliative/supportive care received

SECONDARY OUTCOMES:
Estimation of parameters in the target population associate with cancer-related health care utilization patters including inpatient, emergency room, outpatient visits, lenght of inpatient stay | Patients will be followed from enrolment in the study until death, loss to follow-up, withdrawal of consent or study end date. The minimum follow-up will be 12 months and the maximum allowed follow-up will be 36 months
  * For each health care setting:
    * Number and % of patients with visits
    * Total number of visits
  * Total length of inpatient hospital and ICU stay
Estimation of parameters in the target population associated with treatment- and biopsy-related complications | Patients will be followed from enrolment in the study until death, loss to follow-up, withdrawal of consent or study end date. The minimum follow-up will be 12 months and the maximum allowed follow-up will be 36 months
  * For each treatment complication:
    o Rate of occurrence defined as the number of patients reporting at least one treatment-related complications divided by the number of evaluable patients2 Treatment-related complications can include, but are not limited to nausea and vomiting, diarrhoea, constipation, skin rash, infections, mouth sores, neutropenia, hyponatremia
  * For each biopsy-related complication:
    * Rate of occurrence defined as the number of patients reporting at least one occurrence of the complication divided by the number of patients receiving a biopsy Biopsy-related complications can include but are not limited to collapsed lung, severe bleeding, bronchial spasms, irregular heart rhythms, death, severe chest pain, light-headedness, trouble breathing, excessive bleeding through the bandage, haemoptysis, fever, infection
Estimation of the rate of CNS metastases in the target population including brain metastases and leptomeningeal metastases and treatments associated with CNS metastases | Patients will be followed from enrolment in the study until death, loss to follow-up, withdrawal of consent or study end date. The minimum follow-up will be 12 months and the maximum allowed follow-up will be 36 months
  Overall CNS metastases rate, defined as the number of patients developing CNS metastases divided by the number of evaluable patients
  * Brain metastases rate, defined as the number of patients developing brain metastases divided by the number of evaluable patients
  * Leptomeningeal metastases rate, defined as the number of patients developing leptomeningeal metastases divided by the number of evaluable patients
  * Treatments for CNS metastases, including type of treatment and dates of treatment
Assessment of patient (HRQoL) using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 items (EORTC QLQ-C30) and EORTC QLQ - Lung Cancer 13 items (EORTC QLQ-LC13)3 | Patients will be followed from enrolment in the study until death, loss to follow-up, withdrawal of consent or study end date. The minimum follow-up will be 12 months and the maximum allowed follow-up will be 36 months
  • Change in score from baseline for each Quality of Life (QoL) domain and for overall QoL, measured at each subsequent site visit

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Potter, PhD, MPH, Study Director — AstraZeneca
Locations (110):
- Canada (11):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (8):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Harbin, Heilongjiang
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xian, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Hangzhou, Zhejiang
- France (40):
  - Research Site, Aix-en-Provence, Bouches-du-Rhone
  - Research Site, Brest, Brittany Region
  - Research Site, Tours, Centre-Val de Loire
  - Research Site, Colmar, Haut-Rhin
  - Research Site, Rouen, Haute-Normandie
  - Research Site, Metz-Tessy, Haute-Savoie
  - Research Site, Limoges, Haute-Vienne
  - Research Site, Nantes, Loire-Atlantique
  - Research Site, Saint-Nazaire, Loire-Atlantique
  - Research Site, Angers, Maine-et-Loire
  - Research Site, Lorient, Morbihan
  - Research Site, Saint Priest En Jarez, Pays de la Loire Region
  - Research Site, Marseille, Provence-Alpes-Côte d'Azur Region
  - Research Site, Bayonne, Pyrenees-Atlantiques
  - Research Site, Villefranche-sur-Saône, Rhone
  - Research Site, Le Mans, Sarthe
  - Research Site, Créteil, Val-de-Marne
  - Research Site, Toulon, Var
  - Research Site, Brieuc Cedex 1
  - Research Site, Cannes
  - Research Site, Chambéry
  - Research Site, Clermont-Ferrand
  - Research Site, Gap
  - Research Site, La Réunion
  - Research Site, La Rochelle
  - Research Site, Libourne
  - Research Site, Mantes-la-Jolie
  - Research Site, Meaux
  - Research Site, Montfermeil
  - Research Site, Mulhouse
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Saint-Pierre
  - Research Site, Saint-Quentin
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Troyes
  - Research Site, Suresnes, Île-de-France Region
- Spain (24):
  - Research Site, Seville, Andalusia
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Badalona, Barcelona
  - Research Site, Mataró, Barcelona
  - Research Site, Sabadell, Barcelona
  - Research Site, Jerez de la Frontera, Cadiz
  - Research Site, Las Palmas de Gran Canaria, Canary Islands
  - Research Site, A Coruña, Galicia
  - Research Site, Majadahonda, Madrid
  - Research Site, Pozuelo de Alarcón, Madrid
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Research Site, Reus, Tarragona
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Granada
  - Research Site, Jaén
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Navarra
  - Research Site, Pontevedra
  - Research Site, Seville
  - Research Site, Zaragoza
- Taiwan (8):
  - Research Site, Taichung, Taichung Municipality
  - Research Site, Changhua
  - Research Site, Hsinchu
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- United Kingdom (19):
  - Research Site, Whitchurch, Cardiff
  - Research Site, Hull, East Riding Of Yorkshire
  - Research Site, Brighton, East Sussex
  - Research Site, Maidstone, Kent
  - Research Site, Metropolitan Borough of Wirral, Liverpool
  - Research Site, Birmingham
  - Research Site, Bristol
  - Research Site, Camberley
  - Research Site, Glasgow
  - Research Site, Ipswich
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Nottingham
  - Research Site, Scunthorpe
  - Research Site, Sheffield
  - Research Site, Wolverhampton
  - Research Site, Worcester

IPD SHARING:
Plan to Share IPD: Undecided